CLINICAL TRIAL: NCT02309515
Title: Impact of Short Term Lenalidomide on Immune Response to Prevnar 13® in Individuals With Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Leukemia (SLL), and Monoclonal B Cell Lymphocytosis (MBL)
Brief Title: Lenalidomide in Improving Immune Response to Vaccine Therapy in Patients With Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Monoclonal B Cell Lymphocytosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC138E; NCI-2014-02373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RV-CL-CLL-PI-003938; MC138E (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-06

CONDITIONS: Monoclonal B-Cell Lymphocytosis; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage I Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lenalidomide, pneumococcal 13-valent conjugate vaccine) (Experimental): Patients receive lenalidomide PO QD on days 1-42 and pneumococcal 13-valent conjugate vaccine IM on day 15.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Pneumococcal 13-valent Conjugate Vaccine
- Arm II (pneumococcal 13-valent conjugate vaccine) (Active Comparator): Patients receive pneumococcal 13-valent conjugate vaccine IM on day 15.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pneumococcal 13-valent Conjugate Vaccine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm I (lenalidomide, pneumococcal 13-valent conjugate vaccine)
Biological: Pneumococcal 13-valent Conjugate Vaccine — Given IM
  Other Names: PCV 13; PCV13 Vaccine; Prevnar 13

SUMMARY:
This randomized phase II trial studies how well lenalidomide improves immune response to pneumococcal 13-valent conjugate vaccine in patients with chronic lymphocytic leukemia, small lymphocytic lymphoma, or monoclonal B cell lymphocytosis. Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Lenalidomide may also improve the effectiveness of pneumococcal 13-valent conjugate vaccine that is used to prevent infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of a 6 week course of low dose lenalidomide to improve the proportion of patients with monoclonal B cell lymphocytosis (MBL) and chronic lymphocytic leukemia (CLL) who develop an immune response to pneumococcal vaccination as measured by the proportion of patients with >= 4-fold rise from pre-vaccine (day 15) for >= 2 of the 3 serotypes measured at 28 days post-vaccination by opsonophagocytic activity (OPA) of antibodies from sera.

SECONDARY OBJECTIVES:

I. Evaluate disease status by physical exam and complete blood counts in patients participating in each arm of the study at the time of the 6 week assessment of immune response.

II. Evaluate time to treatment for progressive CLL for patients on each study arm.

III. Evaluate the adverse events profile in each study arm.

TERTIARY OBJECTIVES:

I. To assess the immune response to pneumococcal vaccination as measured by fold-change from pre-vaccine (day 15) to 28 days post-vaccination in OPA geometric mean titers (GMT) of antibodies from sera.

II. To assess the immune response to pneumococcal vaccination as measured by fold-change from pre-vaccine (day 15) to 28 days post-vaccination in quantitative Streptococcus pneumoniae immunoglobulin G (IgG) GMT of antibodies from sera.

III. Evaluate the effect of 6 weeks of low dose lenalidomide on global immune function including T-cell repertoire, T-cell immune synapse, serum immunoglobulin levels, and absolute numbers of T-cell and natural killer (NK) cells.

OUTLINE: Patients are randomized 1 of 2 treatment arms.

ARM I: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-42 and pneumococcal 13-valent conjugate vaccine intramuscularly (IM) on day 15.

ARM II: Patients receive pneumococcal 13-valent conjugate vaccine IM on day 15.

After completion of study treatment, patients are followed up at day 28, and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of:

  1. CLL according to the National Cancer Institute (NCI) criteria
  2. Small lymphocytic lymphoma (SLL) according to the World Health Organization (WHO) criteria
  3. MBL according to the consensus criteria

     * This includes previous documentation of:

       * Biopsy-proven small lymphocytic lymphoma or
       * Diagnosis of CLL or MBL as evidenced by all of the following:

         * Clonal B-cell population in the peripheral blood with immunophenotyping consistent with CLL defined as:

           * The population of lymphocytes share both B-cell antigens (cluster of differentiation [CD]19, CD20 [typically dim expression], or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc)
           * Clonality as evidenced by k (kappa) or lambda light chain expression (typically dim immunoglobulin expression) or other genetic method (e.g. immunoglobulin heavy chain variable [IGHV] analysis) NOTE: splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
         * Patients with a peripheral blood B-cell lymphocyte count of < 5 x 10^9/L and no evidence of lymphadenopathy or organomegaly will be classified as MBL; patients with a peripheral blood B-cell lymphocyte count of < 5 x 10^9/L who have evidence of lymphadenopathy will be classified as SLL; patients with a peripheral blood B-cell lymphocyte count >= 5 x 10^9/L will be considered to have CLL
         * Before diagnosing MBL, CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescence in situ hybridization (FISH) analysis for t(11;14)(IgH/cyclin D 1 [CCND1]) on peripheral blood or tissue biopsy or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy
* CLL or SLL patients only (does not apply to MBL patients): Rai stage 0-1 (both CLL and SLL patients can be staged using the Rai system)
* Patients must not previously have received the Prevnar 13 pneumococcal vaccination; NOTE: previous vaccination with Pneumovax (PCV23) is permitted but must have been at least 365 days prior to registration
* Patients must be previously untreated and must NOT have any of the following indications for chemotherapy:

  * Evidence of progressive marrow failure as manifested by the development of or worsening anemia (=< 11 g/dL) and/or thrombocytopenia (=< 100 x 10^9/L) not due to autoimmune disease
  * Symptomatic or progressive lymphadenopathy, splenomegaly or hepatomegaly
  * One or more of the following disease-related symptoms:

    * Weight loss >= 10% within the previous 6 months
    * Extreme fatigue attributed to CLL
    * Fevers > 100.4 degree Fahrenheit (o^F) for 2 weeks without evidence of infection
    * Drenching night sweats without evidence of infection Note: 1) Prior chemotherapy or monoclonal antibody based therapy for treatment of CLL or SLL will be considered prior therapy; nutraceutical treatments with no established benefit in CLL (such as epigallocatechin gallate or EGCG, found in green tea or other herbal treatments) will not be considered "prior treatment" 2) Prior corticosteroid therapy for an indication other than CLL/SLL will not be considered "prior treatment"; previous use of corticosteroids for treatment of autoimmune complications of CLL/SLL does not constitute prior therapy for CLL/SLL
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 11.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's disease; if total bilirubin is > 1.5 x ULN, a direct bilirubin should be performed and must be < 1.5 mg/dL for Gilbert's to be diagnosed
* Aspartate transaminase (AST) =< 3 x ULN
* Calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* All study participants must be willing to be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS)® program, and be willing and able to comply with the requirements of the REMS® program; NOTE: Actual registration in the Revlimid REMS® program may occur after the patient is randomized since this requirement only applies to patients randomized to Arm A
* Females of reproductive potential must be willing to adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program; NOTE: This requirement only applies to patients randomized to Arm A
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Palpable lymph nodes > 3 cm in maximal dimension
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Any of the following comorbid conditions:

  * New York Heart Association classification III or IV cardiovascular disease
  * Recent myocardial infarction (=< 30 days)
  * Uncontrolled infection
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Other active primary malignancy requiring treatment or limiting survival to =< 2 years prior to registration
* Any radiation therapy =< 28 days prior to registration
* Any major surgery =< 28 days prior to registration
* Current use of corticosteroids; EXCEPTION: low doses of steroids (=< 10 mg of prednisone or equivalent dose of other steroid) used for treatment of nonhematologic medical conditions; NOTE: previous use of corticosteroids is allowed
* Active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment; NOTE: patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation
* History of deep venous thromboses or pulmonary embolism =< 365 days prior to registration
* Co-existent diffuse large B-cell lymphoma (Richter's transformation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait Shanafelt, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine): Patients receive 2.5 mg lenalidomide PO QD on days 1-14 and 5 mg lenalidomide PO QD on days 15-42 and pneumococcal 13-valent conjugate vaccine IM on day 15.
Period: Overall Study
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine)
Started | 5 | 7
Completed | 5 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients that enrolled to treatment are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine) | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Median (Full Range); unit: years] | 62 [58 to 66] | 60 [38 to 71] | 61 [38 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Successful Response
Description: Rate of response to pneumococcal 13-valent conjugate vaccine defined as a four-fold rise from baseline to 28 days after immunization (day 43) for >= 2 of the 3 serotypes studied by OPA of antibodies from sera.
  The proportion of successes will be estimated in each arm by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated in each arm based on the normal approximation.
Time Frame: Day 43
Population: All patients that were registered and assessed for this endpoint are included in this analysis
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine)
Number analyzed (Participants) | 5 | 6
proportion of participants | 0.2 [0.005 to 0.716] | 0.0 [0.0 to 0.46]

2. Secondary Outcome: Disease Status by Physical Exam and Complete Blood Counts
Description: The distribution of disease status will be evaluated in each arm and will be summarized descriptively. Patients will be classified as responders (complete clinical response, incomplete marrow recovery, partial response) vs. non-responders (stable disease, progressive disease [PD]). For MBL, patients will be classified as not PD vs PD. Differences in disease status response will be compared between the two arms using Fisher's exact test.
Time Frame: At 6 weeks
Population: All patients that registered and were assessed for response were included in this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine)
Number analyzed (Participants) | 5 | 6
Participants
  Responder | 1 | 0
  Non-responder | 4 | 6

3. Secondary Outcome: Incidence of Adverse Events Using NCI Common Terminology Criteria for Adverse Events Version 4.0
Description: Adverse Events were collected during treatment according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse event will be recorded for each patient. The worst grade per patient is presented below.
Time Frame: Up to day 50
Population: All patients that received protocol treatment are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine)
Number analyzed (Participants) | 5 | 6
Participants
  Grade 0 | 2 | 3
  Grade 1 | 3 | 3
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

4. Secondary Outcome: Time to Treatment for Progressive CLL
Description: The distribution of time to treatment will be estimated in each arm using the method of Kaplan-Meier. Time to treatment will be compared between the two arms using log-rank statistics.
Time Frame: Time from the date of registration to the date of initiation of treatment for progressive CLL assessed up to 2 years
Population: The study was terminated prior to the collection of any subsequent treatment for CLL. Therefore, no patients were eligible for this endpoint and this analysis was not performed.
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during one 50 day cycle of treatment.
Description: Adverse events were collected during one 50 day cycle of treatment.
Arm/Group | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) | Arm II (Pneumococcal 13-valent Conjugate Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lenalidomide, Pneumococcal 13-valent Conjugate Vaccine) (N=5) | Arm II (Pneumococcal 13-valent Conjugate Vaccine) (N=6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5)
Fatigue (General disorders) | 2 (3) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 2 (4)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT02309515/Prot_SAP_000.pdf